CLINICAL TRIAL: NCT05493137
Title: Investigating Physical Activity Levels of Parents of Children With Cystic Fibrosis and Its Influence on Their Children's Physical Activity Levels and Nebuliser Use
Brief Title: Physical Activity Levels of Parents of Children With Cystic Fibrosis- (PHACTS-CF)
Acronym: PHACTS-CF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Kieren Lock, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A096376
Record Dates: First submitted 2022-08-04; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Cystic Fibrosis in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention will be provided — No intervention will be provided, this is an observational study

SUMMARY:
This study will investigate if parental physical activity levels, assessed by providing a physical activity questionnaire to parents of children aged 6-16 with Cystic Fibrosis (CF), is associated with their child with CF's physical activity levels. Children's activity levels will be taken from electronic records where a questionnaire is routinely given at annual reviews to analyse this. Parental activity levels will also be compared against adherence to nebulisers as a proxy for adherence to treatment, this data is again in the electronic records of patients and is collected at annual reviews.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of Children aged 5-16 years.
2. Under the care of Cambridge University Hospitals CF team
3. Confirmed Cystic Fibrosis diagnosis
4. Uses an ineb as main nebulizer delivery device.
5. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Parents of CYP diagnosed with a CF screen positive inconclusive diagnosis (SPID).
2. If not yet doing lung function.
3. If has any other self-identified physical disability which may limit physical activity.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents of children with cystic fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
GPAQ | Reviews the past 7 days activities.
  Activity questionnaire for parents

SECONDARY OUTCOMES:
CPAQ | Reviews the past 7 days activities.
  Physical activity Questionnaire for children aged 5-11 (From medical notes)
YPAQ | Reviews the past 7 days activities.
  Physical activity Questionnaire for children aged 12 and over (From medical notes)
Ineb adherence | 1 year
  Adherence to recommended number of nebulised treatment from the i-adhere software downloaded from the ineb device.
Lung function | Best score in the last 1 year.
  FEV1 (z-score and %), FVC (z-score and %), FEF2575 (z-score and %) (From medical notes)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.